CLINICAL TRIAL: NCT04689659
Title: Multi-centers, Open-Label, Phase 2 Study to Evaluate the Efficacy and Safety of Donor-Derived CD7 CAR T Cells in Subjects With Relapsed or Refractory T-cell Leukemia/Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-IIT-LCYJ-2020-005
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: T-cell Leukemia/Lymphoma; Refractory T Lymphoblastic Leukemia/Lymphoma; Relapse/Recurrence
Keywords: CAR-T
MeSH Terms: conditions — Leukemia, T-Cell; Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- chimeric antigen receptor T cell treatment (Experimental)
  Interventions: Biological: chimeric antigen receptor T cell treatment

INTERVENTIONS:
Biological: chimeric antigen receptor T cell treatment — CD7 CAR T cells will be given once intravenously at one dose (1×106, with an allowance of ± 20%) in patients received previous HSCT donor-derived CAR T cells. Patients who received fresh donor derived CD7 CAR T cells were given initial dose of 1×106, with an allowance of ± 20%. The dose levels may be adjusted during the study based on the specific number of cells on the day of fresh CAR T cells infusion, due to at this time all the patients have completed lymphodepleting, so we adopt the allowance of ±20% for each group of absolute infusion cells. And patients who were lower than the designed dose group were also given infusion, but they will be either assigned to the lower dose group or exclude from safety analysis of designed dose group.

SUMMARY:
This is a multi-centers, single-arm, open label, Phase 2 clinical trial to evaluate the efficacy and safety of CD7 CAR T cells in subjects with relapsed or refractory T-cell leukemia/lymphoma. Seventy subjects will be enrolled. CD7 CAR T cells will be given once intravenously at one dose (1×106, with an allowance of ± 20%) in patients received previous HSCT donor-derived CAR T cells. Patients who received fresh donor derived CD7 CAR T cells were given initial dose of 1×106, with an allowance of ± 20%. The dose levels may be adjusted during the study based on the specific number of cells on the day of fresh CAR T cells infusion, due to at this time all the patients have completed lymphodepleting, so we adopt the allowance of ±20% for each group of absolute infusion cells. And patients who were lower than the designed dose group were also given infusion, but they will be either assigned to the lower dose group or exclude from safety analysis of designed dose group.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Candidates with relapse or refractory CD7+ T cell acute lymphoblastic leukemia/lymphoma, who have progressed on after treatment with all standard therapies or intolerant of standard care, have limited prognosis with currently available therapies and had no available curative treatment options (such as SCT or chemotherapy)
2. Male or female, aged 1-70 years
3. No serious allergic constitution
4. Eastern Cooperative Oncology Group (ECOG) performance status (Oken et al., 1982) score 0 to 2
5. Have life expectancy of at least 60 days based on investigator's judgement
6. CD7 positive in bone marrow or cerebrospinal fluid (CSF) by flow cytometry, or CD7 positive in tumor tissues by immunohistochemistry; (CD7 positive criteria: Flow cytometry: Positive: > 80% of tumor cells expressed CD7 and the mean fluorescence (MFI) of CD7 is the same as that in normal T cells; Dim: > 80% of tumor cells expressed CD7, but the MFI of CD7 is lower than that in normal T cells as least as 1log; Partial positive: 20-80% of tumor cells expressed CD7 and the MFI of CD7 is the same as that in normal T cells. tumor tissue immunohistochemistry: Positive > 30% tumor cells expressed CD7);
7. Provide a signed informed consent before any screening procedure; subjects who voluntarily participate in the study should have the ability to understand and sign the informed consent form and be willing to follow the study visit schedule and relevant study procedure, as specified in the protocol. Candidates aged 19-70 years need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form; Children candidates of 1-7 can be recruited after the legal guardian or patient advocate has signed the treatment consent form and voluntary consent form. Children candidates of 8-18 years old need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form and their legal guardian or patient advocate has also need to sign the treatment consent form and voluntary consent form, respectively

Exclusion criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Intracranial hypertension or disorder of consciousness
2. Symptomatic heart failure or severe arrhythmia
3. Symptoms of severe respiratory failure
4. Complicated with other types of malignant tumors
5. Diffuse intravascular coagulation
6. Serum creatinine and / or blood urea nitrogen ≥ 1.5 times of the normal value
7. Suffering from septicemia or other uncontrollable infections
8. Patients with uncontrollable diabetes
9. Severe mental disorders
10. Obvious and active intracranial lesions were detected by cranial magnetic resonance imaging (MRI)
11. Have received organ transplantation (excluding bone marrow transplant)
12. Reproductive-aged female patients with positive blood human chorionic gonadotropin (HCG) test
13. Screened to be positive of infection of hepatitis (including hepatitis B and C), acquired immunodeficiency syndrome (AIDS) or syphilis

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: Best overall response (BOR) rate | at 3 months
  Best overall response (BOR) rate to the CAR T treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan J, Zhao L, Zhang Y, Seery S, Tan Y, Deng B, Shan L, Ling Z, Wu F, Wang Z, Wang Q, Yu X, Zheng Q, Xu X, Yuan Y, Tian Z, Zhang Y, Peng S, Chang AH, Feng X. Donor-derived CD7 CAR T cells for pediatric and adult relapsed/refractory T-ALL/LBL: a phase 2 trial. Blood. 2025 Dec 4;146(23):2745-2757. doi: 10.1182/blood.2025029299. PMID 40712157
- [Derived] Velasquez MP. Allogeneic CD7-CAR T cells to bridge the gap? Transplant Cell Ther. 2023 Mar;29(3):139-140. doi: 10.1016/j.jtct.2023.02.006. No abstract available. PMID 36858787
- [Derived] Pan J, Tan Y, Wang G, Deng B, Ling Z, Song W, Seery S, Zhang Y, Peng S, Xu J, Duan J, Wang Z, Yu X, Zheng Q, Xu X, Yuan Y, Yan F, Tian Z, Tang K, Zhang J, Chang AH, Feng X. Donor-Derived CD7 Chimeric Antigen Receptor T Cells for T-Cell Acute Lymphoblastic Leukemia: First-in-Human, Phase I Trial. J Clin Oncol. 2021 Oct 20;39(30):3340-3351. doi: 10.1200/JCO.21.00389. Epub 2021 Jul 29. PMID 34324392